CLINICAL TRIAL: NCT01193699
Title: An Open-label, Prospective, Multicentre, Phase I/II Dose Escalation Study to Determine the Maximum Tolerated Dose and to Assess the Safety and Efficacy of P1101, PEG-Proline-Interferon Alpha-2b in Patients With Polycythaemia Vera
Brief Title: Safety Study of Pegylated Interferon Alpha 2b to Treat Polycythemia Vera
Acronym: PEGINVERA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P11012010
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P1101 (Experimental)
  Interventions: Drug: PEG-P-INF alpha-2b (P1101)

INTERVENTIONS:
Drug: PEG-P-INF alpha-2b (P1101) — µg (starting with 50 µg), subcutaneously, 2-weekly administration

SUMMARY:
The purpose of this study is the identification of the maximum tolerated dose (MTD) of the investigational medicinal product. Moreover the safety and tolerability will be assessed and an exploratory analysis of efficacy and biomarker modulation will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study specific screening activities and able to comply with this protocol.
2. Patients age ≥18 years
3. Confirmed diagnosis of PV according to either the WHO criteria (2008, appendix 6) or the PSVG (appendix 7) criteria plus JAK-2 positivity, including newly diagnosed, pre-treated and on cytoreductive therapy.
4. Eastern Cooperative Oncology Group performance status ≤ 2
5. If female of childbearing potential - have a negative urine pregnancy test result within 7 days prior to the scheduled first application of investigational product and agree to employ adequate birth control measures for the duration of the study.

Exclusion criteria:

1. Diagnosis of any other myeloproliferative disorder
2. Any clinically significant illness or surgery within 4 weeks prior to dosing
3. Systemic infections, e.g. hepatitis B, hepatitis C, or HIV at screening
4. Uncontrolled hypertension (systolic > 150 mmHg and diastolic > 100 mmHg, or clinically significant (i.e. active) cardiovascular disease: CVA/stroke (≤ 3 months prior to enrolment), myocardial infarction (≤ 3 months prior to enrolment), significant coronary artery stenosis, unstable angina, New York Heart Association (NYHA) Class 2 or greater Congestive heart failure, or serious cardiac arrhythmia requiring medication.
5. Previous treatment with Interferon for PV
6. Concurrent treatment with cytoreductive agents other than Hydroxyurea and investigational agents of any type
7. History of malignant disease, including solid tumours and haematological malignancies (except basal cell and squamous cell carcinomas of the skin and carcinoma in situ of the cervix that have been completely excised and are considered cured) within the last 3 years
8. History of severe allergic (like anaphylaxis) or hypersensitivity reactions (like angioedema), any known or suspected intolerance to the investigational product.
9. Use of any investigational drug or participation in any investigational drug study within the last 4 weeks
10. Clinically significant history or known presence of psychiatric disorders, including but not limited to depression, anxiety and sleep disorders
11. Organ transplant, past or planned
12. Inadequate liver function defined by serum (total) bilirubin > 2,5 x ULN and/ or AST and ALT > 2,5 x ULN
13. Clinically significant ECG findings
14. History of renal disease requiring haemodialysis or seizure disorder requiring anticonvulsant therapy
15. Pregnant or lactating females (pregnancy test to be assessed within 7 days prior to study treatment start)
16. Acute or chronic infections or autoimmune diseases (collagen diseases, polyarthritis, immune thrombocythemia, thyroiditis, psoriasis, lupus nephritis or any other autoimmune disorder).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-08 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | The incidence of dose limiting toxicities (DLTs), which define the MTD are assessed continously until achievement of MTD.
  The definition of MTD is based on a 3+3 dose escalation design. MTD is defined as the next lower dose of that dose which was considered to be untolerated (observed DLT frequency at least 2 out of 3 in one cohort or at least 2 out of six patients in 2 cohorts).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grohmann-Izay, MD, Study Director — AOP Orphan Pharmaceuticals AG
Locations (4):
- Austria (4):
  - Innsbruck, Tyrol
  - Wels, Upper Austria
  - Salzburg
  - Vienna

REFERENCES:
- [Derived] Gisslinger H, Zagrijtschuk O, Buxhofer-Ausch V, Thaler J, Schloegl E, Gastl GA, Wolf D, Kralovics R, Gisslinger B, Strecker K, Egle A, Melchardt T, Burgstaller S, Willenbacher E, Schalling M, Them NC, Kadlecova P, Klade C, Greil R. Ropeginterferon alfa-2b, a novel IFNalpha-2b, induces high response rates with low toxicity in patients with polycythemia vera. Blood. 2015 Oct 8;126(15):1762-9. doi: 10.1182/blood-2015-04-637280. Epub 2015 Aug 10. PMID 26261238